CLINICAL TRIAL: NCT06287905
Title: A Comparative Study of Using Scorpion Antivenom Versus Scorpion Antivenom and Prazosin Drug for Scorpion Stings Management in Sohag University Hospitals
Brief Title: A Comparative Study of Using Scorpion Antivenom Versus Scorpion Antivenom and Prazosin
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Meray Medhat Shokry, lecturer of clinical toxicology, Sohag University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-23-02-24
Record Dates: First submitted 2024-02-19; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Morality
Keywords: mortality, scorpion, antivenom, prazosin
MeSH Terms: interventions — Prazosin

STUDY DESIGN:
Intervention Model Description: observational comparative
Who Masked: Participant
Masking Description: Simple randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group of antivenom only (No Intervention): Dose of antivenom 1-1 ampoule intramuscular and/ or, 2-1 to 5 Polyvalent anti-scorpion serum ampoules produced by the vaccine & serum institution (VACSERA)in Egypt according to the severity of the case on 200 to 500 ml glucose 5% infusion and assess the patient clinically to repeat the dose after 4 to 6 hours. (Shoreit et al., 2019)
- group of adding prazosin plus standard treatment (Experimental): 1-Dose and administration of prazosin: 30 μg/kg/dose of prazosin will be delivered orally every 6 hours 4 doses, in adults we shouldn't exceed 1 mg per dose. Prazosin will be delivered using a nasogastric tube while securing the patient's airway in the event of vomiting or unconsciousness. Every 30 minutes for the first three hours, every hour for the following six, and then every four hours until improvement, blood pressure, pulse rate, respiration rate, and oxygen saturation will be measured. When pain is the only symptom, prophylaxis shouldn't be given. To avoid the first-dose phenomenon, the patient should remain in a laying position for around 3 hours (even while the case is being examined) (Shoreit et al., 2019).
  Interventions: Drug: Prazosin Oral Tablet

INTERVENTIONS:
Drug: Prazosin Oral Tablet — 1-Dose and administration of prazosin: 30 μg/kg/dose of prazosin will be delivered orally every 6 hours 4 doses, in adults we shouldn't exceed 1 mg per dose. Prazosin will be delivered using a nasogastric tube while securing the patient's airway in the event of vomiting or unconsciousness. Every 30 minutes for the first three hours, every hour for the following six, and then every four hours until improvement, blood pressure, pulse rate, respiration rate, and oxygen saturation will be measured. When pain is the only symptom, prophylaxis shouldn't be given. To avoid the first-dose phenomenon, the patient should remain in a laying position for around 3 hours (even while the case is being examined) (Shoreit et al., 2019).
  Arms: group of adding prazosin plus standard treatment

SUMMARY:
Interventional study designed for the evaluation of characters and the outcome of scorpion sting patients will admit to Sohag University Hospitals in 2 randomized groups. The first group will receive scorpion antivenom only whether by the intravenous or the intramuscular route of administration. The second group will receive a combination of prazosin plus scorpion antivenom whether by the intravenous or the intramuscular route of administration. Both groups will receive proper first aid and supportive treatment

DETAILED DESCRIPTION:
Tools of the study:

1. Dose and administration of prazosin: 30 μg/kg/dose of prazosin will be delivered orally every 6 hours 4 doses, in adults we shouldn't exceed 1 mg per dose. Prazosin will be delivered using a nasogastric tube while securing the patient's airway in the event of vomiting or unconsciousness. Every 30 minutes for the first three hours, every hour for the following six, and then every four hours until improvement, blood pressure, pulse rate, respiration rate, and oxygen saturation will be measured. When pain is the only symptom, prophylaxis shouldn't be given. To avoid the first-dose phenomenon, the patient should remain in a laying position for around 3 hours (even while the case is being examined) (Shoreit et al., 2019).

   Dose of antivenom 1-1 ampoule intramuscular and/ or, 2-1 to 5 Polyvalent anti-scorpion serum ampoules produced by the vaccine & serum institution (VACSERA)in Egypt according to the severity of the case on 200 to 500 ml glucose 5% infusion and assess the patient clinically to repeat the dose after 4 to 6 hours. (Shoreit et al., 2019)
2. A prepared sheet containing

   1. the demographic characteristics of each patient
   2. Vital signs and degree of coma at time of admission of the patient.
   3. First aid management as resuscitation.
   4. Supportive management will be done to the patients during the admission will be recorded.
   5. Cardiac enzymes measurements, duration of hospital stay and the outcome of patients in each group.

ELIGIBILITY:
Inclusion criteria:

* History and clinical diagnosis of scorpion sting
* Admit in Sohag University hospitals
* During the period from February 2023 to July 2024.
* Accepting informed written consent from the case itself or the first degree relative if the case will underage or in a coma.

Exclusion Criteria:

* .All other envenomation cases or poisoning will be excluded.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | "up to 1 month"
  record the mortality rate in the two groups during the hospital stay

SECONDARY OUTCOMES:
Morbidity | "through the study completion an average of a 1 year "
  assess any complications with the patients in the two groups fever, allergy, hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Meray M Shokry Zaghary, Principal Investigator — Sohag University
Locations (1):
- Meray Medhat Shokry Zaghary, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No